CLINICAL TRIAL: NCT00319644
Title: Impact of Using Mini-Bronchoalveolar Lavage as a Diagnostic Test for Ventilator-Associated Pneumonia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 27831-01
Record Dates: First submitted 2006-04-27; First posted 2006-04-27 (Estimated); Results first posted 2012-11-16 (Estimated); Last update posted 2012-11-16 (Estimated); Status verified 2012-10

CONDITIONS: Ventilator-Associated Pneumonia
MeSH Terms: conditions — Pneumonia, Ventilator-Associated | interventions — Bronchoalveolar Lavage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Minibal Arm (Experimental): Using Mini bronchoalveolar lavage
  Interventions: Device: Bronchoalveolar lavage
- Tracheal Aspirates (No Intervention): standard of care for ICU.

INTERVENTIONS:
Device: Bronchoalveolar lavage — Using catheter to obtain respiratory sample
  Other Names: MiniBal
  Arms: Minibal Arm

SUMMARY:
The proposed study will evaluate adult patients admitted to the medical or surgical intensive care units (ICUs) at San Francisco General Hospital (SFGH). On admission, patients will be randomized in a 1:1 manner to the mini-bronchoalveolar lavage (BAL) quantitative culture arm in the setting of suspected ventilator-associated pneumonia (VAP) versus the tracheal aspirate culture arm, which is the current test available at SFGH.

DETAILED DESCRIPTION:
Patients will be randomized to either Mini-Bal or tracheal aspirate then samples will be taken to the lab for culture. Comparative analysis will then be performed based upon lab results.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (> age 18) admitted to 5E, 5R, and 4E intensive care units and are on the ventilator for greater than 48 hours and expected to remain on the ventilator for awhile
* Study procedures would be performed only in patients clinically suspected of having VAP.

Exclusion Criteria:

* Severe respiratory distress at the time of suspected VAP defined by:

  * FiO2 ≥ 0.7
  * PEEP ≥ 12

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2006-05; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julin F Tang, M.D., M.S., Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco General Hospital, San Francisco, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was a randomized, controlled trial of adult patients admitted to the trauma/surgical intensive care unit of San Francisco General Hospital and was conducted from 5/1/2005 to August 15, 2008
Pre-assignment Details: Adult patients with suspected VAP were randomized to the mini-BAL (MB) diagnostic group or the tracheal aspirate (TA) diagnostic group.
Groups:
- Tracheal Aspirates: No intervention. Standard of care in ICU.
Period: Overall Study
Arm/Group | Tracheal Aspirates | Minibal Arm
Started | 21 | 16
Completed | 21 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Minibal Arm | Tracheal Aspirates | Total
Number analyzed (Participants) | 16 | 21 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 21 | 37
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 49.38 (16.3) | 52.81 (19.3) | 51.09 (27.45)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 10 | 12
  Male | 14 | 11 | 25
Region of Enrollment [Number; unit: participants]
  United States | 16 | 21 | 37

OUTCOME MEASURES:

1. Primary Outcome: Change in Antibiotic Usage or Exposure
Description: We expect that 100-110 adult patients will have clinically suspected VAP over a 2-year period. We assume that 50 patients with suspected VAP will be randomized to mini-BAl, and 50 patients will be randomized to tracheal aspirate. We expect that patients randomized to tracheal aspirate group will receive an average of approximately 14 total days of antibiotics over their ICU stay. This study will have >80% power to detect a difference of 4 days of antibiotics (i.e. average of 10 days in mini-BAL group) with a 7-day standard deviation in both groups (alpha error level 5%).
Time Frame: It is theorized that patients randomized to the tracheal aspirate will receive an average of 15 days of antibiotics while patients randomized under the minibal arm will receive an average of 10 days of antibiotics
Population: Of the 37 adult critically ill patients, 21 belonged to the tracheal aspirate (TA) group and 16 patients were classified as mini-BAL (MB) group.
Measure: Mean (Standard Deviation); unit: days
Groups:
- Mini-BAL: BAL for quantitative culture as TA group.
- Tracheal Aspirates: No intervention. Standard of care in ICU. the aspirates were sent for micro culture.
Arm/Group | Mini-BAL | Tracheal Aspirates
Number analyzed (Participants) | 16 | 21
days | 11.87 (13.80) | 7.76 (1.06)
Statistical Analysis 1: Comparison: Mini-BAL vs Tracheal Aspirates; The chi-square test(or Fisher exact test where needed) was used to compare proportions with dichotomous variables. The Student-t test was used for quantitative variables woth normal distribution, and Mann-Whitney-U test was used for data not normally distributed; Test type: Superiority or Other; p = 0.26, Chi-squared; Mean Difference (Final Values) = 20

2. Primary Outcome: Antibiotics Exposure Days
Description: We hypothesize that Mini-BAL quantitative culture in place of tracheal aspirate culture will reduce the total days of antibiotics exposure
Time Frame: 15 days
Population: Random
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Mini-BAL | Tracheal Aspirates
Number analyzed (Participants) | 16 | 21
days | 4 (3.89) | 5.81 (6.95)

ADVERSE EVENTS:
Arm/Group | Minibal Arm | Tracheal Aspirates
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/21
Other Adverse Events (participants affected / at risk) | 2/16 | 0/21
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Minibal Arm (N=16) | Tracheal Aspirates (N=21)
Transient Desaturation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No